CLINICAL TRIAL: NCT00789022
Title: Glutamatergic Amino Acids and Oxytocin Levels in the Plasma of Patients in First Psychotic Episode (FPE)- Before and After Neuroleptic Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Dr. Uri Nitzan, Resident
Other Study IDs: uriel111
Record Dates: First submitted 2008-11-09; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Schizophrenia; Schizophreniform; Schizoaffective Disorder; Brief Psychotic Episode
Keywords: First-Psychotic-Episode (FPE); Glutamatergic system; Glycine; D-Serine; Oxytocin; Estrogen
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 40 subjects in a First Psychotic Episode
- 2: 20 First Degree relatives
- 3: 20 Healthy subjects

SUMMARY:
The goal of our research is to check the levels of D-Serine, Glycine, and other Glutamatergic amino acids, in patients with First Psychotic Episode (FPE). These patients are in the early stage of the disease, treated with neuroleptics for short periods of time, and are usually hospitalized for the first time. The hypothesis of the research is that we will find low levels of Glycine and D-Serine in these patients. Following an Anti-psychotic treatment we will expect these levels to return to the norm, and that this correction will be accompanied by a reduction of positive and negative symptoms.

In addition, we will check the D-Serine and Glycine levels in the plasma of first degree relatives of the patients and a group of healthy subjects. The results of this study might support the hypothesis that the Glutamatergic system in involved in the pathology of Schizophrenia from it's early stages.

In addition, we will check the levels of Oxytocin and Estrogen in the plasma of patients in FPE. Our hypothesis is that we will find low levels of Estrogen and High levels of Oxytocin in this group of patients. The results of the study might support the hypothesis that Estrogen and Oxytocin are involved in the pathology of Schizophrenia from it's early stages.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18-60 years
* Clinical Diagnosis of Schizophrenia, Schizophreniphorm disorder, Schizoaffective Disorder, Brief esychotic episode

Exclusion Criteria:

* two years or more of positive symptoms
* Neuroleptic treatment for more then twe weeks in the prior month, or for more then six weeks at any time.
* Drug induced psychotic episode

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hospitalized patients First degree ralatives Healthy subjects from the community
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Glycine and D-Serine levels in the plasma. | 6-8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Medical Center, Hod Hasharom, Israel